CLINICAL TRIAL: NCT04898426
Title: Effect of Enhanced Interactive Text Messages and Phone Instruction on the Quality of Bowel Preparation for Colonoscopy: a Randomised Controlled Trial.
Brief Title: Effect of Enhanced Interactive Text Messages and Phone Instruction on the Quality of Bowel Preparation for Colonoscopy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Griffith Base Hospital (Other)
Responsible Party: Principal Investigator, Dr Minh Pham, Researcher, Griffith Base Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: GriffithBH
Record Dates: First submitted 2021-05-11; First posted 2021-05-24 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Colon Polyp; Colon Neoplasm
Keywords: Colonoscopy; Boston bowel preparation scale; Bowel preparation quality; Enhanced bowel preparation instruction
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient cannot be blinded to the allocation. The colonoscopist (care provider) is blinded to the allocation. The investigator and statistician will remain blinded to the allocation until analysis has been conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Bowel Preparation Instruction (No Intervention): Patients receive the standard-of-care bowel preparation instruction.
- Enhanced Bowel Preparation Instruction (Experimental): Patients receive enhanced instructions (SMS, phone call, info website) in addition to the standard-of-care bowel preparation instruction.
  Interventions: Other: Enhanced bowel preparation instruction

INTERVENTIONS:
Other: Enhanced bowel preparation instruction — Automated delivery of SMS, pre-recorded phone call, and link to an information website.
  Arms: Enhanced Bowel Preparation Instruction

SUMMARY:
Efficacy Evaluation of Enhanced Bowel Preparation Instructions in Elective Colonoscopy.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled clinical investigation designed to evaluate the efficacy of enhanced bowel preparation instructions (automated SMS, information website, and pre-recorded phone call) in improving bowel preparation quality in elective colonoscopy.

Subjects from the interventional and control group will receive standard of care bowel preparation instruction.

The interventional group will receive enhanced instructions delivered by automated SMS, information website and pre-recorded phone calls in the 48 hours leading up to the colonoscopy day. The intention is to provide a reminder, to reiterate instruction on clear fluid diet and timing of bowel preparation medication, and to provide additional graphical illustration on the information website.

Subjects in the interventional group must reply "OK" to each automated SMS or press "1" on the keypad at the end of the automated phone call to acknowledge understanding and receipt of instruction. Failure to acknowledge trigger an alert for a booking office staff member to directly call the patient and confirm compliance.

The clinical investigation will be conducted at one hospital in the state of New South Wales, Australia.

Subjects will be randomized to the interventional group (enhanced instruction) versus the control group (standard instruction).

The proceduralist assessing outcome measures at the time of colonoscopy is blinded to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Elective colonoscopy booking at Griffith Base Hospital.

Exclusion Criteria:

* Emergency colonoscopy
* Patients who are unable to understand bowel preparation instructions in the following languages: English, Italian, Punjabi, Gujarati, Samoan, Mandarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Bowel preparation quality | Bowel preparation quality is scored once for each patient at the time of colonoscopy completion. We expect to conduct this score in 500 patients over the study period of approximately 12 months.
  Bowel preparation quality is assessed using the Boston Bowel Preparation Scale (range 0 to 9, with higher scores indicating better bowel preparation quality)

SECONDARY OUTCOMES:
Colonoscopy cancellation rate | Colonoscopy cancellation rate will be calculated at the time of study completion, expected to be 12 months.
  The number of colonoscopy being cancelled within 48 hours of the colonoscopy date. The rates will be compared between the study groups.
Caecal intubation rate | Caecal intubation rate will be calculated at the time of study completion, expected to be 12 months.
  The proportion of colonoscopies in which the colonoscope reaches the furthest extent of the colon. The rates will be compared between the study groups.
Polyp detection rate | Polyp detection rate will be calculated at the time of study completion, expected to be 12 months.
  The proportion of colonoscopies in which a polyp was detected. The rates will be compared between the study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Minh Pham, Principal Investigator — Researcher
Locations (1):
- Griffith Base Hospital, Griffith, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rex DK, Imperiale TF, Latinovich DR, Bratcher LL. Impact of bowel preparation on efficiency and cost of colonoscopy. Am J Gastroenterol. 2002 Jul;97(7):1696-700. doi: 10.1111/j.1572-0241.2002.05827.x. PMID 12135020
- [Background] Chokshi RV, Hovis CE, Hollander T, Early DS, Wang JS. Prevalence of missed adenomas in patients with inadequate bowel preparation on screening colonoscopy. Gastrointest Endosc. 2012 Jun;75(6):1197-203. doi: 10.1016/j.gie.2012.01.005. Epub 2012 Feb 28. PMID 22381531
- [Background] Froehlich F, Wietlisbach V, Gonvers JJ, Burnand B, Vader JP. Impact of colonic cleansing on quality and diagnostic yield of colonoscopy: the European Panel of Appropriateness of Gastrointestinal Endoscopy European multicenter study. Gastrointest Endosc. 2005 Mar;61(3):378-84. doi: 10.1016/s0016-5107(04)02776-2. PMID 15758907
- [Background] Harewood GC, Sharma VK, de Garmo P. Impact of colonoscopy preparation quality on detection of suspected colonic neoplasia. Gastrointest Endosc. 2003 Jul;58(1):76-9. doi: 10.1067/mge.2003.294. PMID 12838225
- [Background] Guo X, Yang Z, Zhao L, Leung F, Luo H, Kang X, Li X, Jia H, Yang S, Tao Q, Pan Y, Guo X. Enhanced instructions improve the quality of bowel preparation for colonoscopy: a meta-analysis of randomized controlled trials. Gastrointest Endosc. 2017 Jan;85(1):90-97.e6. doi: 10.1016/j.gie.2016.05.012. Epub 2016 May 14. PMID 27189659
- [Background] Kang X, Zhao L, Leung F, Luo H, Wang L, Wu J, Guo X, Wang X, Zhang L, Hui N, Tao Q, Jia H, Liu Z, Chen Z, Liu J, Wu K, Fan D, Pan Y, Guo X. Delivery of Instructions via Mobile Social Media App Increases Quality of Bowel Preparation. Clin Gastroenterol Hepatol. 2016 Mar;14(3):429-435.e3. doi: 10.1016/j.cgh.2015.09.038. Epub 2015 Oct 20. PMID 26492848
- [Background] Liu X, Luo H, Zhang L, Leung FW, Liu Z, Wang X, Huang R, Hui N, Wu K, Fan D, Pan Y, Guo X. Telephone-based re-education on the day before colonoscopy improves the quality of bowel preparation and the polyp detection rate: a prospective, colonoscopist-blinded, randomised, controlled study. Gut. 2014 Jan;63(1):125-30. doi: 10.1136/gutjnl-2012-304292. Epub 2013 Mar 16. PMID 23503044
- [Background] Lee YJ, Kim ES, Choi JH, Lee KI, Park KS, Cho KB, Jang BK, Chung WJ, Hwang JS. Impact of reinforced education by telephone and short message service on the quality of bowel preparation: a randomized controlled study. Endoscopy. 2015 Nov;47(11):1018-27. doi: 10.1055/s-0034-1392406. Epub 2015 Jul 16. PMID 26182387
- [Background] Spiegel BM, Talley J, Shekelle P, Agarwal N, Snyder B, Bolus R, Kurzbard N, Chan M, Ho A, Kaneshiro M, Cordasco K, Cohen H. Development and validation of a novel patient educational booklet to enhance colonoscopy preparation. Am J Gastroenterol. 2011 May;106(5):875-83. doi: 10.1038/ajg.2011.75. Epub 2011 Apr 12. PMID 21483463
- [Background] Calderwood AH, Lai EJ, Fix OK, Jacobson BC. An endoscopist-blinded, randomized, controlled trial of a simple visual aid to improve bowel preparation for screening colonoscopy. Gastrointest Endosc. 2011 Feb;73(2):307-14. doi: 10.1016/j.gie.2010.10.013. Epub 2010 Dec 18. PMID 21168840
- [Background] Janahiraman S, Tay CY, Lee JM, Lim WL, Khiew CH, Ishak I, Onn ZY, Ibrahim MR, Chew CK. Effect of an intensive patient educational programme on the quality of bowel preparation for colonoscopy: a single-blind randomised controlled trial. BMJ Open Gastroenterol. 2020 May;7(1):e000376. doi: 10.1136/bmjgast-2020-000376. PMID 32371502
- [Background] Walter B, Frank R, Ludwig L, Dikopoulos N, Mayr M, Neu B, Mayer B, Hann A, Meier B, Caca K, Seufferlein T, Meining A. Smartphone Application to Reinforce Education Increases High-Quality Preparation for Colorectal Cancer Screening Colonoscopies in a Randomized Trial. Clin Gastroenterol Hepatol. 2021 Feb;19(2):331-338.e5. doi: 10.1016/j.cgh.2020.03.051. Epub 2020 Mar 30. PMID 32240835